CLINICAL TRIAL: NCT02319967
Title: Coordinated Healthcare Interventions for Childhood Asthma Gaps in Outcomes (CHICAGO Plan)
Brief Title: Coordinated Healthcare Interventions for Childhood Asthma Gaps in Outcomes
Acronym: CHICAGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Sinai Health System (Other); Cook County Health & Hospitals System (Other); Rush University Medical Center (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); University of Chicago (Other); Chicago Department of Public Health (Other Government); Respiratory Health Association (Unknown); Chicago Asthma Consortium (Unknown); Illinois Institute of Technology (Other); Illinois Emergency Department Asthma Surveillance Project (Unknown); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jerry Krishnan, Associate Vice Chancellor for Population Health Sciences, Professor of Medicine and Public Health, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-1214; AS-1307-05420 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2014-12-15; First posted 2014-12-19 (Estimated); Results first posted 2019-04-22 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Asthma
Keywords: community health worker; emergency; asthma
MeSH Terms: conditions — Asthma; Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced usual care (No Intervention): Inhaler technique education and distribution of spacers to all participants.
- ED-only (Experimental): Inhaler technique education and distribution of spacers to all participants. Structured patient-centered ED discharge template (CAPE) to be completed by ED coordinator.
  Interventions: Behavioral: CAPE
- ED-plus-home (Experimental): Inhaler technique education and distribution of spacers to all participants. Structured patient-centered ED discharge template (CAPE) to be completed by ED coordinator.
  Home visits by a community health worker (CHW).
  Interventions: Behavioral: CAPE; Behavioral: CHW home visits

INTERVENTIONS:
Behavioral: CAPE — Decision support and communication tool to promote guideline-recommended care by providers and use of such care by children/caregivers
  Arms: ED-only; ED-plus-home
Behavioral: CHW home visits — Home visits by community health workers (CHW) to assist children and their caregivers to implement the CAPE and other guideline-recommended competencies.
  Arms: ED-plus-home

SUMMARY:
Chicago is an epicenter for asthma health disparities in the U.S., with African-American children 5-11 yrs bearing a disproportionate share of the burden. Among the most visible of these disparities is the high rate of visits to the Emergency Department (ED) for uncontrolled asthma. Clinical uncertainties regarding the real-world effectiveness of guideline recommendations for ED discharge and strategies to reduce environmental triggers at home contribute to practice variation and poor adherence to guidelines. The CHICAGO Plan tests both ED- and home-level interventions to improve clinically meaningful outcomes in a minority pediatric ED population with uncontrolled asthma.

ELIGIBILITY:
Inclusion criteria (all of the following):

1. Child is 5-11 years of age (a population in whom a diagnosis of asthma is generally reliable, and in whom exacerbations are common);
2. Child is presenting to the ED, urgent care center, or observation unit at a participating clinical center (Anne and Robert H. Lurie Children's Hospital of Chicago, Sinai Health System's Mount Sinai Hospital, John H. Stroger Jr. Hospital of Cook County Health & Hospitals System, Rush University Medical Center, University of Chicago Medicine Comer Children's Hospital, and the University of Illinois Hospital & Health Sciences System);
3. Child is treated with at least 1 dose of an inhaled or nebulized short-acting bronchodilator (quick-relief medication);
4. Child received systemic corticosteroids in the ED OR the caregiver reported at least 1 additional acute care visit for asthma in the previous 6 months (defined as an asthma-related ED visit or urgent care visit, or course of systemic corticosteroids);
5. Child and caregiver approached at least 1 hour after receipt of the first dose of quick-relief medication or systemic corticosteroids, whichever occurred first;
6. Diagnosis of asthma exacerbation by treating clinician;
7. Treating ED clinician indicates the child is likely to be discharged to home; and
8. Caregiver reports that English or Spanish is the preferred language at home.

Exclusion criteria (none of the following):

1. Caregiver declines to provide informed consent, or the child declines to provide assent;
2. Child is admitted to an intensive care unit or transferred to another healthcare facility;
3. Child or another member of the child's primary household is a current or previous participant in the CHICAGO Plan;
4. Child is enrolled in another study involving a health-related intervention;
5. A CHW is already visiting the home as part of another program;
6. Child does not reside in Chicago.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 373 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry A Krishnan, MD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (6):
- United States (6):
  - Sinai Health System, Chicago, Illinois
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Cook County Health & Hospitals System, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois

REFERENCES:
- [Derived] Krishnan JA, Martin MA, Lohff C, Mosnaim GS, Margellos-Anast H, DeLisa JA, McMahon K, Erwin K, Zun LS, Berbaum ML, McDermott M, Bracken NE, Kumar R, Margaret Paik S, Nyenhuis SM, Ignoffo S, Press VG, Pittsenbarger ZE, Thompson TM; CHICAGO Plan consortium. Design of a pragmatic trial in minority children presenting to the emergency department with uncontrolled asthma: The CHICAGO Plan. Contemp Clin Trials. 2017 Jun;57:10-22. doi: 10.1016/j.cct.2017.03.015. Epub 2017 Mar 31. PMID 28366780
- See also: Patient-Centered Outcomes Research Institute (PCORI): Funding award details — http://www.pcori.org/research-results/2013/coordinated-healthcare-interventions-childhood-asthma-gaps-outcomes-chicago

RESULTS

PARTICIPANT FLOW:
Groups:
- ED-only: Inhaler technique education and distribution of spacers to all participants. Structured patient-centered ED discharge template (CAPE) to be completed by ED coordinator.
  CAPE: Structured patient-centered ED discharge template completed prior to ED discharge.
- ED-plus-home: Inhaler technique education and distribution of spacers to all participants. Structured patient-centered ED discharge template (CAPE) to be completed by ED coordinator.
  Community-health worker-led home visits.
  CAPE: Structured patient-centered ED discharge template completed prior to ED discharge.
  Home: Home visits led by community-health workers to reinforce CAPE and guide environmental remediation.
Period: Overall Study
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Started | 126 | 126 | 121
Completed | 78 | 82 | 76
Not Completed | 48 | 44 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home | Total
Number analyzed (Participants) | 126 | 126 | 121 | 373
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.3 (1.9) | 7.4 (2.0) | 7.3 (1.9) | 7.4 (1.9)
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorial: 5-7 years | 72 | 75 | 70 | 217
  Age, Categorial: 8-11 years | 54 | 51 | 51 | 156
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 35 | 42 | 124
  Male | 79 | 91 | 79 | 249
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 37 | 41 | 116
  Not Hispanic or Latino | 87 | 87 | 80 | 254
  Unknown or Not Reported | 1 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 3 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 81 | 81 | 77 | 239
  White | 39 | 38 | 38 | 115
  More than one race | 2 | 7 | 5 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: PROMIS Asthma Impact Scale (v1.0, SF8a)
Description: Raw scores (0-32) were converted to T-scores to measure change from index visit to 6-month primary endpoint. Low scores indicate better asthma; high scores indicate worse asthma.
  PROMIS Asthma Impact Scale, Pediatric: Min possible T-score: 31.5; Max possible T-score: 76.2 Possible range for change in T-score is [-44.7 to 44.7]
  PROMIS Asthma Impact Scale, Parent proxy: Min possible T-score: 32; Max possible T-score: 80 Possible range for change in T-score is [-48 to 48]
  The reported value represents a change in T-score from baseline to 6 months after index ED discharge.
  A negative change in score indicates improvement in asthma. A positive change in score indicates worsening of asthma. A score of 0 indicates no change.
Time Frame: Baseline and 6 months after index ED discharge
Population: The number of participants analyzed refers to the number of participants with evaluable data at baseline and 6 months after index ED discharge. The number of participants included in the analysis may not match the total number of participants enrolled as we were unable to obtain outcome data from some participants.
Measure: Median (Inter-Quartile Range); unit: T-score
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Number analyzed (Participants) | 78 | 82 | 76
T-score | -7.8 [-17.3 to 0.0] | -9.3 [-16.4 to -5.0] | -11.9 [-19.3 to -6.0]

2. Primary Outcome: PROMIS Satisfaction With Participation in Social Roles (v1.0, SF4a)
Description: Raw scores (4-20) were converted to T-scores to measure change from index visit to 6-month primary endpoint. Low scores indicate less satisfaction among caregivers; high scores indicate more satisfaction among caregivers.
  PROMIS Satisfaction With Participation in Social Roles: Min possible T-score: 29.0; Max possible T-score: 64.1 Possible range for change in T-score is [-35.1 to 35.1]
  The reported value represents a change in T-score from baseline to 6 months after index ED discharge.
  A negative change in score indicates less satisfaction among caregivers. A positive change in score indicates a more satisfaction among caregivers. A score of 0 indicates no change.
Time Frame: Baseline and 6 months after index ED discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T-score
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Number analyzed (Participants) | 76 | 82 | 75
T-score | 0.0 [-6.0 to 6.1] | 0.0 [-3.5 to 9.7] | 0.0 [-4.3 to 6.8]

3. Secondary Outcome: Childhood Asthma Control Test (cACT)
Description: The scores of each item were summed for a total score (0-27) to measure change from index to 6-month primary endpoint. Low scores indicate worse asthma; high scores indicate better asthma.
  Childhood Asthma Control Test (cACT): Min possible score: 0; Max possible score: 27 Possible range for change in score is [-27 to 27]
  The reported value represents a change in score from baseline to 6 months after index ED discharge.
  A negative change in score indicates improvement in asthma. A positive change in score indicates worsening of asthma. A score of 0 indicates no change.
Time Frame: Baseline and 6 months after index ED discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Number analyzed (Participants) | 33 | 34 | 24
score | 3.0 [1.0 to 6.0] | 4.0 [1.2 to 5.8] | 5.5 [3.0 to 7.2]

4. Secondary Outcome: PROMIS Anxiety (v1.0, SF4a)
Description: Raw scores (4-20) were converted to T-scores to measure change from index visit to 6-month primary endpoint. Low scores indicate less anxiety; high scores indicate more anxiety.
  PROMIS Anxiety: Min possible T-score: 40.3; Max possible T-score: 81.6 Possible range for change in T-score is [-41.3 to 41.3]
  The reported value represents a change in T-score from baseline to 6 months after index ED discharge.
  A negative change in score indicates improvement in anxiety. A positive change in score indicates worsening of anxiety. A score of 0 indicates no change.
Time Frame: Baseline and 6 months after index ED discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T-score
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Number analyzed (Participants) | 66 | 80 | 67
T-score | -3.2 [-10.9 to 0.0] | -3.8 [-11.2 to 0.0] | -2.5 [-13.4 to 1.9]

5. Secondary Outcome: PROMIS Depression (v1.0, SF4a)
Description: Raw scores (4-20) were converted to T-scores to measure change from index visit to 6-month primary endpoint. Low scores indicate less depression; high scores indicate more depression.
  PROMIS Depression: Min possible T-score: 41.0; Max possible T-score: 79.4 Possible range for change in T-score is [-38.4 to 38.4]
  The reported value represents a change in T-score from baseline to 6 months after index ED discharge.
  A negative change in score indicates improvement in depression. A positive change in score indicates worsening of depression. A score of 0 indicates no change.
Time Frame: Baseline and 6 months after index ED discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T-score
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Number analyzed (Participants) | 67 | 79 | 68
T-score | 0.0 [-2.2 to 0.0] | 0.0 [-4.9 to 0.0] | 0.0 [-7.3 to 0.0]

6. Secondary Outcome: PROMIS Fatigue (v1.0, SF4a)
Description: Raw scores (4-20) were converted to T-scores to measure change from index visit to 6-month primary endpoint. Low scores indicate less fatigue; high scores indicate more fatigue.
  PROMIS Fatigue: Min possible T-score: 33.7; Max possible T-score: 75.8 Possible range for change in T-score is [-42.1 to 42.1]
  The reported value represents a change in T-score from baseline to 6 months after index ED discharge.
  A negative change in score indicates improvement in fatigue (i.e., less fatigue). A positive change in score indicates worsening of fatigue (i.e., more fatigue). A score of 0 indicates no change.
Time Frame: Baseline and 6 months after index ED discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T-score
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Number analyzed (Participants) | 64 | 79 | 67
T-score | 0.0 [-9.4 to 8.2] | 0.0 [-8.5 to 4.4] | -2.6 [-12.2 to 1.4]

7. Secondary Outcome: PROMIS Sleep Disturbance (v1.0, SF4a)
Description: Raw scores (4-20) were converted to T-scores to measure change from index visit to 6-month primary endpoint. Low scores indicate less sleep disturbance; high scores indicate more sleep disturbance.
  PROMIS Sleep Disturbance (v1.0, SF4a): Min possible T-score: 32.0; Max possible T-score: 73.3 Possible range for change in T-score is [-41.3 to 41.3]
  The reported value represents a change in T-score from baseline to 6 months after index ED discharge.
  A negative change in score indicates improvement in sleep disturbance (i.e., less sleep disturbance). A positive change in score indicates worsening of sleep disturbance (i.e., more sleep disturbance). A score of 0 indicates no change.
Time Frame: Baseline and 6 months after index ED discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T-score
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Number analyzed (Participants) | 64 | 77 | 65
T-score | 0.0 [-4.1 to 4.0] | 0.0 [-3.7 to 2.4] | -1.9 [-4.0 to 2.4]

8. Secondary Outcome: Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ)
Description: The overall score is the mean score across all 13 items. Each item is scored on a 7-point Likert scale with 1 indicating severe impairment and 7 indicating no impairment. Higher scores indicate better quality of life; lower scores indicate worse quality of life.
  Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ): Min possible score: 1; Max possible score: 7 Possible range for change in score is [-6 to 6]
  The reported value represents a change in overall score from baseline to 6 months after index ED discharge.
  A negative change in score indicates worsening quality of life. A positive change in score indicates improvement in quality of life. A score of 0 indicates no change.
Time Frame: Baseline and 6 months after index ED discharge
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Number analyzed (Participants) | 63 | 74 | 64
score | 0.8 [0.0 to 2.1] | 1.1 [0.1 to 2.2] | 1.2 [0.2 to 2.2]

9. Secondary Outcome: Number of Participants With All-cause Emergency Department (ED) or Urgent Care Visits
Description: Count of participants (children) with at least one all-cause ED or urgent care visit at 6 months
Time Frame: 6 months post index ED discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Number analyzed (Participants) | 126 | 126 | 121
Participants | 54 | 53 | 44

10. Secondary Outcome: Number of Participants With All-cause Hospitalizations
Description: Count of participants (children) with at least one all-cause hospitalization at 6 months
Time Frame: 6 months post index ED discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Number analyzed (Participants) | 126 | 126 | 121
Participants | 12 | 11 | 9

11. Secondary Outcome: Self-management Practices After ED Discharge: Number of Participants Who Filled Prescriptions for Systemic Corticosteroids
Description: Count of participants who filled a prescription for systemic corticosteroids within 7 days of discharge
Time Frame: 7 days post index ED discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Number analyzed (Participants) | 100 | 108 | 97
Participants | 82 | 89 | 79

12. Secondary Outcome: Self-management Practices After ED Discharge: Number of Participants Who Filled Prescriptions for Inhaled Corticosteroids or Other Controller
Description: Count of participants who filled prescription for inhaled corticosteroids or other controller within 7 days of discharge
Time Frame: 7 days post index ED discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Number analyzed (Participants) | 100 | 108 | 97
Participants | 42 | 49 | 69

13. Secondary Outcome: Self-management Practices After ED Discharge: Number of Participants Who Attended an Outpatient Appointment With Patient-identified Asthma Provider
Description: Count of participants who attended follow-up appointment with patient-identifier asthma provider within 4 weeks of discharge
Time Frame: 4 weeks post index ED discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Number analyzed (Participants) | 115 | 114 | 111
Participants | 37 | 48 | 57

14. Secondary Outcome: Indicator of Guideline-consistent Care Provided on ED Discharge: Number of Participants Who Received Instructions to Use Systemic Corticosteroids
Description: Count of participants who were provided documented discharge instructions to use systemic corticosteroids
Time Frame: At index ED discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Number analyzed (Participants) | 126 | 126 | 121
Participants | 77 | 125 | 118

15. Secondary Outcome: Indicator of Guideline-consistent Care Provided on ED Discharge: Number of Participants Who Received Instructions to Use Inhaled Corticosteroids or Other Controller
Description: Count of participants who were provided documented discharge instructions to use inhaled corticosteroids or other controller
Time Frame: At index ED discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Number analyzed (Participants) | 126 | 126 | 121
Participants | 52 | 80 | 87

16. Secondary Outcome: Indicator of Guideline-consistent Care Provided on ED Discharge: Number of Participants Who Received Instructions to Use Inhaled Rescue Medication
Description: Count of participants who were provided documented discharge instructions to use an inhaled rescue medication
Time Frame: At index ED discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Number analyzed (Participants) | 126 | 126 | 121
Participants | 107 | 125 | 118

17. Secondary Outcome: Indicator of Guideline-consistent Care Provided on ED Discharge: Number of Participants Who Received a Follow-up Appointment Scheduled by ED Staff
Description: Count of participants who were provided documented discharge instructions for a follow-up appointment scheduled within 4 weeks of discharge
Time Frame: At index ED discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care | ED-only | ED-plus-home
Number analyzed (Participants) | 126 | 126 | 121
Participants | 10 | 62 | 56

ADVERSE EVENTS:
Time Frame: 6 months
Description: Participants were recruited in the emergency department during an asthma exacerbation. As reviewed and approved by the study's independent data and safety monitoring board, subsequent visits to the emergency department and hospitalizations were expected in this population and were, therefore, not reported as serious adverse events or other adverse events.
Groups:
- Usual Care: Inhaler technique education and distribution of spacers to all participants.
- CAPE: Inhaler technique education and distribution of spacers to all participants. Structured patient-centered ED discharge template (CAPE) to be completed by ED coordinator.
  CAPE: Structured patient-centered ED discharge template completed prior to ED discharge.
- CAPE + Home: Inhaler technique education and distribution of spacers to all participants. Structured patient-centered ED discharge template (CAPE) to be completed by ED coordinator.
  Community-health worker-led home visits.
  CAPE: Structured patient-centered ED discharge template completed prior to ED discharge.
  Home: Home visits led by community-health workers to reinforce CAPE and guide environmental remediation.
Arm/Group | Usual Care | CAPE | CAPE + Home
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/126 | 0/121
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/126 | 0/121
Other Adverse Events (participants affected / at risk) | 0/126 | 0/126 | 0/121

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT02319967/Prot_SAP_000.pdf